CLINICAL TRIAL: NCT01454297
Title: A Prospective, Longitudinal, Observational Study in Newly Diagnosed Multiple Myeloma (MM) Patients to Assess the Relationship Between Patient Outcomes, Treatment Regimens and Molecular Profiles
Brief Title: Relating Clinical Outcomes in Multiple Myeloma to Personal Assessment of Genetic Profile
Acronym: CoMMpass
Status: Completed | Type: Observational
Sponsor: Multiple Myeloma Research Foundation (Other)
Collaborators: Translational Genomics Research Institute (Other); Corewell Health West (Other); Van Andel Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: MMRF-11-001
Record Dates: First submitted 2011-10-07; First posted 2011-10-19 (Estimated); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Multiple Myeloma
Keywords: Myeloma; Multiple Myeloma; Observational; Longitudinal
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bone marrow, Peripheral Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Newly diagnosed Multiple Myeloma: This is a prospective observational study in patients with symptomatic multiple myeloma who have not yet initiated therapy for their disease.

SUMMARY:
The primary objective of this observational study is to identify the molecular profiles and clinical characteristics that define subsets of myeloma patients during the course of the disease.

DETAILED DESCRIPTION:
Understanding the molecular basis of cancer is a critical step toward devising the most effective treatment of the patient as an individual. The promise of molecular targeted therapeutics and personalized cancer care has been demonstrated in breast and lung cancer and chronic myeloid leukemia. However, similar examples of success in multiple myeloma have not been achieved despite extensive basic research as well as clinical advances. What is well understood is that myeloma is a heterogeneous disease with great genetic and epigenetic complexity.22, 23 Therefore, there remains a critical need to understand myeloma patient biology in the context of current patient care.24 The objective of this longitudinal study is to identify patient subgroups and phenotypes defined by molecular profiling and clinical features. These profiles will enable a better understanding of mechanisms of disease, drug response and patient relapse. Ultimately the study is intended to drive successful drug development and patient care in multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years old.
* Patient has been diagnosed with symptomatic MM with measurable disease that includes at least one of the following:

Serum M protein ≥ 1g/dl Urine M protein ≥ 200 mg/24 hrs Involved free light chain level ≥ 10 mg/dl and an abnormal serum free light chain ratio (<0.26 or >1.65).

* The patient is a candidate for systemic therapy that includes an IMiD® (e.g., lenalidomide, pomalidomide, thalidomide) and/or proteasome inhibitor (e.g., bortezomib, carfilzomib) as part of the initial regimen.
* No more than 30 days from baseline bone marrow evaluation as per this protocol to initiation of first-line therapy.
* Patient has read, understood and signed informed consent.

Exclusion Criteria:

* Patient is already receiving systemic therapy for MM (a single dose of bisphosphonates and up to 100 mg total dose of dexamethasone or equivalent corticosteroids are permitted prior to registration on study).
* Patient had another malignancy within the last 5 years (except for basal or squamous cell carcinoma, or in situ cancer of the cervix).
* Patient is enrolled in a blinded clinical trial for the first-line treatment of multiple myeloma. Patients may be enrolled in subsequent clinical trials as long as continued access to data and tissue, as per this protocol, is not prohibited.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed, symptomatic, multiple myeloma, candidates for systemic treatment
Sampling Method: Non-Probability Sample
Enrollment: 1154 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Molecular profiles and clinical characteristics that define subsets of myeloma patients at initial diagnosis and at relapse of disease. | Baseline to 8 years.
  Standard clinical and laboratory assessments. Genomic tests (DNA and RNA sequencing, etc.) on bone marrow aspirates obtained at baseline, suspected complete response, and relapse/progression.

SECONDARY OUTCOMES:
Response rates | Up to one year after baseline.
  IMWG criteria: stringent complete response, complete response, very good partial response, partial response, no response.
Survival rates | Five to eight years after baseline
  Progression-free survival and overall survival
Bone disease assessed radiographically | Baseline and during five to eight years of follow-up
Health-related quality of life | Baseline and during five to eight years of follow-up
  EORTC QLQ-C30 and QLQ-MY20
Resource utilization | Baseline and during five to eight years of follow-up
  Hospitalizations and ER visits
Severe adverse events | Five to eight years
  Severe/CTCAE grade 3-4 adverse events (checklist)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Auclair, Study Director — Multiple Myeloma Research Foundation
Locations (73):
- United States (55):
  - Mayo Clinic Campus in Scottsdale, AZ, Scottsdale, Arizona
  - UC San Diego Moores Cancer Center, San Diego, California
  - Sharp Health Care, San Diego, California
  - VA San Diego Healthcare System, San Diego, California
  - San Francisco VA Medical Center, San Francisco, California
  - UCSF Medical Center, San Francisco, California
  - Kaiser Permanente of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Carl and Dorothy Bennett Cancer Center, Stamford, Connecticut
  - VA Medical Center, Washington DC,, Washington D.C., District of Columbia
  - Ocala Oncology Center, Ocala, Florida
  - Winship Cancer Institute - Emory University, Atlanta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - University of Chicago, Chicago, Illinois
  - Illinois Cancer Specialists, Niles, Illinois
  - Cancer Center of Kansas, Wichita, Kansas
  - Peninsula Regional Cancer Center, Salisbury, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Mayo Clinic-Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Kansas City VA Medical Center, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - Billings Clinic, Billings, Montana
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Broome Oncology, Johnson City, New York
  - New York University Medical Center, New York, New York
  - Mt Sinai Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College-NY Presbyterian Hospital, New York, New York
  - St Francis Hospital, Roslyn, New York
  - Eastchester Center for Cancer Care, The Bronx, New York
  - Waverly Hematology Oncology, Cary, North Carolina
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - First Health Outpatient Cancer Center, Pinehurst, North Carolina
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Northwest Cancer Specialists, PC, Tualatin, Oregon
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Baylor Research Institute, Dallas, Texas
  - University of Texas Southwest Medical Center, Dallas, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - Central Texas VA Healthcare Center, Temple, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Texas Oncology- Waco, Waco, Texas
  - Virginia Cancer Specialists PV, Fairfax, Virginia
  - Cancer Care Northwest, Spokane, Washington
  - Yakima Valley Memorial Hospital/North Star Lodge, Yakima, Washington
  - Marshfield Clinic, Marshfield, Wisconsin
- Canada (4):
  - Tom Baker Cancer Centre, Alberta Health Services, Calgary, Alberta
  - Cross Cancer Institute, Alberta Health Services, Edmonton, Alberta
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - McGill University Health Center, Royal Victoria Hospital, Montreal, Quebec
- Spain (14):
  - Hospital Clinica Universitari Lozano Blesa, Zaragoza, Aragon
  - Hospital Univ Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Son Llàtze, Palma de Mallorca, Balearic Islands
  - Hospital University de Salamanca, Salamanca, Castille and León
  - H. U. Germans Trias i Pujol, Badalona, Catalonia
  - Hospital Quirón de Madrid, Pozuelo de Alarcón, Madrid
  - University Hospital Infanta Sofia, San Sebastián de los Reyes, Madrid
  - Clínica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Universitari de Canarias, Santa Cruz de Tenerife, Santa Cruz
  - Hospital del Mar, Barcelona
  - Hospital Santa Creu I Sant Pau, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital Ramón y Cajal, Madrid
  - Hospital Puerta de Hierro, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Interim Analysis data will be released every 6 months

REFERENCES:
- [Derived] Auclair D, Mansfield C, Fiala MA, Chari A, Cole CE, Kaufman JL, Orloff GJ, Siegel DS, Zonder JA, Mange B, Yesil J, Dalal M, Mikhael JR. Preferences and Priorities for Relapsed Multiple Myeloma Treatments Among Patients and Caregivers in the United States. Patient Prefer Adherence. 2022 Mar 1;16:573-585. doi: 10.2147/PPA.S345906. eCollection 2022. PMID 35256844
- [Derived] Barwick BG, Gupta VA, Matulis SM, Patton JC, Powell DR, Gu Y, Jaye DL, Conneely KN, Lin YC, Hofmeister CC, Nooka AK, Keats JJ, Lonial S, Vertino PM, Boise LH. Chromatin Accessibility Identifies Regulatory Elements Predictive of Gene Expression and Disease Outcome in Multiple Myeloma. Clin Cancer Res. 2021 Jun 1;27(11):3178-3189. doi: 10.1158/1078-0432.CCR-20-2931. Epub 2021 Mar 17. PMID 33731366
- [Derived] Foltz SM, Gao Q, Yoon CJ, Sun H, Yao L, Li Y, Jayasinghe RG, Cao S, King J, Kohnen DR, Fiala MA, Ding L, Vij R. Evolution and structure of clinically relevant gene fusions in multiple myeloma. Nat Commun. 2020 May 29;11(1):2666. doi: 10.1038/s41467-020-16434-y. PMID 32471990
- [Derived] Miller A, Asmann Y, Cattaneo L, Braggio E, Keats J, Auclair D, Lonial S; MMRF CoMMpass Network; Russell SJ, Stewart AK. High somatic mutation and neoantigen burden are correlated with decreased progression-free survival in multiple myeloma. Blood Cancer J. 2017 Sep 22;7(9):e612. doi: 10.1038/bcj.2017.94. PMID 28937974
- See also: The Multiple Myeloma Research Foundation — http://www.themmrf.org